CLINICAL TRIAL: NCT04266704
Title: Building a Multidisciplinary Research Program to Address Hypertension Disparities: Exploring the Neurocognitive Mechanisms of a Self-Management Intervention for African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lenette M. Jones, Assistant professor, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00226482; 1K01HL145366-01 (NIH)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Along with providing education on a low sodium diet (Dietary Approaches to Stop Hypertension or DASH), exercise, and medication adherence, the intervention arm is designed to promote information sharing and stimulate broad cortical neural networks, the default mode (DMN), which focuses on emotion-management and self-awareness.
  Interventions: Behavioral: Sharing Intervention
- Control (Active Comparator): education on a low sodium diet (Dietary Approaches to Stop Hypertension or DASH), exercise, and medication adherence
  Interventions: Behavioral: Sharing Intervention

INTERVENTIONS:
Behavioral: Sharing Intervention — intervention includes both analytic and socioemotional components related to self-management of hypertension and is specifically targeted to African American women. Along with providing education on lifestyle changes to lower blood pressure, DASH diet, exercise, and medication adherence (analytic components), the intervention is designed to promote social activities around blood pressure self-management, in particular, sharing blood pressure management information with peers (socioemotional components).

SUMMARY:
The goal of this project is to develop and pilot test a research protocol to assess the influence of a health information behavior enhanced intervention on self-management, blood pressure control, and brain activity in African American women with hypertension. This work will identify characteristics of African American women that are associated with improved self-management and decreased blood pressure, and subsequent reduction of risk of heart disease and premature death. The results of this project will have direct impact in informing interventions to improve blood pressure control, by advancing our knowledge of brain activity associated with behavior change in African American women with hypertension in the metro-Detroit area, and ultimately everywhere.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria are (a) aged >18, (b) clinically diagnosed with hypertension, and (c) right-handed (due to potential differences in brain morphology compared to left-handed individuals).

-

Exclusion Criteria: Exclusion criteria are (a) history of renal insufficiency, (b) score less than 22 on the Montreal Cognitive Assessment (MOCA), and (c) having one of the following contraindications for fMRI: heart pacemaker, heart defibrillator, metal in the eye, and some types of metal elsewhere within the body such as certain surgical clips for aneurysms in the head, heart valve prostheses, electrodes, and some other implanted devices, pregnant. We require a score of >22 on the MOCA to assure that subjects are able to participate cognitive procedures.

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — African American women
Enrollment: 50 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Brain activity | 6 months
  ability to differentiate between analytic and empathetic prompts, subset of sample

SECONDARY OUTCOMES:
Blood pressure | Baseline and 6 months
  Systolic and diastolic
Quality of life-PROMIS | Baseline and 6 months
  Quality of life - PROMIS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No